CLINICAL TRIAL: NCT06081543
Title: A Prospective Randomized Unblinded Study of Ketogenetic Versus Mixed Diet on Exercise Tolerance in Subjects With the Metabolic Phenotype of Heart Failure With Preserved Ejection Fraction
Brief Title: Ketogenic Diet vs Mixed Diet in Patients With Heart Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Yuchi Han, Professor-Clinical, Cardiovascular Medicine, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2022H0366; CDMRP-PR212399-E (Other Grant/Funding Number: Departent of Defense)
Record Dates: First submitted 2023-09-26; First posted 2023-10-13 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: Ketogenic Diet; Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketogenic Diet (Experimental): This arm will be provided food to induce a state of nutritional ketosis in each person as defined as blood Beta-hydroxybutyrate (3-OHB) ≥0.5 millimoles (mM), which will require most participants to consume <50 g/day carbohydrate and 1.5g/kg reference weight protein. Fat will comprise the remaining calories with an emphasis on monounsaturated and saturated sources from whole foods.
  Interventions: Dietary Supplement: Ketogenic diet
- Low-fat mixed Diet (Experimental): This arm will be provided food consisting of ~25% fat, and the remaining calories from carbohydrate (~55% after accounting for protein at ~20%).
  Interventions: Dietary Supplement: Low-fat Mixed diet

INTERVENTIONS:
Dietary Supplement: Ketogenic diet — Participants will undertake a controlled feeding intervention. All food will be prepared and delivered to participants by research staff for the first 6 weeks. After that will be a free-living diet period where food will not be supplied but participants will receive educational materials and frequent coaching from a dietitian to help maintain the specified diet. Participants will be asked to exclusively follow the diet in efforts to control any dietary effects.
  Arms: Ketogenic Diet
Dietary Supplement: Low-fat Mixed diet — Participants will undertake a controlled feeding intervention. All food will be prepared and delivered to participants by research staff for the first 6 weeks. After that will be a free-living diet period where food will not be supplied but participants will receive educational materials and frequent coaching from a dietitian to help maintain the specified diet. Participants will be asked to exclusively follow the diet in efforts to control any dietary effects.
  Arms: Low-fat mixed Diet

SUMMARY:
This study is being done to evaluate the effects of a low carbohydrate ketogenic diet (KD) versus a low-fat diet (MD) on exercise tolerance in participants with heart failure with normal pumping function and diabetes or pre-diabetes, or metabolic syndrome, or obesity.

DETAILED DESCRIPTION:
Participants will be randomized to either a ketogenic diet (KD), or a low-fat diet (MD).

Participants will eat the specified diet for a period of 6-months and be supported by dietary coaching. All foods and/or groceries will be provided at no cost for the first six weeks of the study.

After the initial 6 weeks, and for the next 20-22 weeks, participants will change into a free-living diet period where food will not be supplied but they will receive educational materials and frequent coaching from a dietitian to help maintain the specified diet. Both diets are based on a slight reduction in dietary caloric requirements, so some weight loss should occur over the 6-month intervention.

Ketone and glucose values will be monitored over a 2-week period at baseline, during the conclusion of the first 6 weeks, as well as the final 2-week period at the end of the 6-month study. Participants will apply a sensor one week prior to starting the study to capture one week of baseline metabolic status and the first week of the diet. Another sensor will be applied for week 5 to week 7, and a third sensor for weeks 25 to 26 at the end of the diet. Weight, blood pressure, oxygen saturation, resting heart rate, and activity level will also be monitored.

Throughout the duration of the study, participants will be monitored closely, and diabetes and diuretics medications adjusted by physicians involved in this study. Other medications will be continued and guided by your regular physicians. Both groups will be supported from the research physicians on a weekly basis (including medication changes). The duration of the study is expected to last for approximately 6-month.

All participants will undergo the following tests on 2 separate visit days at these 3 testing time points during the study (baseline, 6 weeks, and end of the study (26 weeks) unless specified.

These tests include:

1. An in-person physical exam by one of the physician investigators.
2. A Dual-energy X-ray absorptiometry (DXA) test, which is a test to measure your body composition. There is a small amount of radiation used in DXA, which is extremely low (by comparison, a standard chest x-ray is 125 times more radiation than a DXA scan).
3. Two cardiac magnetic resonance imaging (MRI) scans. One consisting of non-contrast resting scans including elastography (MR safe drum-like device will generate mechanical waves on specific organs to test the stiffness of these organs) and another consisting of a contrast-enhanced MRI scan of the heart (The one with contrast will only be performed twice for the study, once at the baseline and once end of the study).
4. A six-minute walk test (6MWT). You will walk along an even, undisturbed corridor for 6 minutes. A qualified person will supervise your test. The test has been used as a measure of exercise capacity in many patient populations and is extremely safe.
5. A cardiopulmonary stress test (CPET), also know as an oxygen consumption test (VO2). During the CPET you will be asked to exercise on a treadmill or using an ergometer while breathing into a mask. This will be performed on a separate day from the 6MWT.
6. Up to four tablespoons of blood will be drawn for a number of tests. Blood draws may cause discomfort at the skin puncture site and a small bruise may develop that may persist for several weeks. There is also a small possibility of an infection. These risks are identical to standard clinical blood draws.
7. A 24-hour urine collection.

ELIGIBILITY:
Inclusions:

1. Age ≥ 18 years old and ≤ 80 years old & willingness to be randomized to either diet.
2. NYHA class I - III for at least 3 months.
3. Ejection fraction ≥40% by biplane 2D, or 3D echo, or CMR
4. Echo findings of abnormal or indeterminant diastolic function or right heart catheterization (RHC) data: At rest: mean pulmonary capillary wedge pressure (PCWP) > 15 mmHg. pulmonary vascular resistance (PVR) < 3 Wood Units.
5. Stable medical therapy for at least 3 months as determined by the treating physician (no new cardiac or diabetic medications within 3 months of enrollment or during enrollment and dosage should be stable for 1 month prior to enrollment).
6. Dose of oral diuretics changes allowed but must be stable for 1 week prior to randomization.
7. Body Mass Index (BMI) ≥ 25 or Type 2 Diabetes Mellitus or prediabetes (fasting glucose of 100 - 125 mg/dL or glycated hemoglobin (A1C) 5.7-6.4% or metabolic syndrome.
8. Ability to participate in exercise treadmill testing.
9. Ability to sign written consent.

Exclusions:

1. Women who are pregnant, current breast-feeding, or have intention to become pregnant while in the study.
2. Known allergy or sensitivity to gadolinium-based contrast agents.
3. Implanted pacemaker, cardioverter defibrillator, Cardiac resynchronization therapy, left ventricular assist device.
4. Other metallic implants/aneurysm clips that are contraindicated in MRI.
5. Claustrophobia
6. History of severe kidney disease of estimated glomerular filtration rate (eGFR) <30 ml/kg/1.73m2.
7. Type I diabetes.
8. History of diabetic ketoacidosis.
9. Prior diagnosis of oxygen dependent pulmonary disease.
10. Body Mass Index (BMI) < 25.
11. Recent acute myocardial infarction or acute coronary syndrome (30 days).
12. Or recent (within 30 days) or planned (within 30 days) cardiac revascularization History of left main disease, severe triple vessel disease, coronary artery bypass graft surgery.
13. Left ventricular ejection fraction < 50%.
14. Uncontrolled systemic systolic blood pressure (SBP)/diastolic blood pressure (DBP) hypertension (SBP >180 or DBP >110 mmHg).
15. Severe stenotic or regurgitant valvular heart disease, expected to lead to surgery during the study period.
16. Persistent atrial fibrillation.
17. History of uncontrolled or untreated ventricular arrhythmias.
18. Cardiovascular diseases or treatments that increase the unpredictability of or change the subject's clinical course, independent of heart failure.
19. Heart transplant or listing for heart transplant.
20. Cardiomyopathy based on infiltrative diseases (e.g. amyloidosis), accumulation diseases (e.g. haemochromatosis, Fabry disease), muscular dystrophies, cardiomyopathy with reversible causes (e.g. stress cardiomyopathy), hypertrophic obstructive cardiomyopathy or known pericardial constriction.
21. Acute decompensated heart failure requiring intravenous diuretics, vasodilators, inotropic agents or mechanical support within 1 week of screening and during the screening period prior to randomization.
22. Hemoglobin of <9 g/dL at screening.
23. Major surgery (major according to the investigator's assessment) performed within 90 days prior to screening, or major scheduled elective surgery (e.g. hip replacement) within 90 days after screening.
24. Acute or chronic liver disease, defined by serum levels of transaminases or alkaline phosphatase more than three times the upper limit of normal at screening.
25. Gastrointestinal surgery or gastrointestinal disorder that might interfere with diet. Prior bariatric surgery allowed if weight-stable for past 3 months.
26. Any documented active or suspected malignancy or history of malignancy within 2 years prior to screening, except appropriately treated basal cell carcinoma of the skin, in situ carcinoma of the uterine cervix, or low-risk prostate cancer (subjects with pre-treatment prostate-specific antigen levels of <10 ng/mL, and biopsy Gleason scores of ≤6 and clinical stage T1c or T2a).
27. Presence of any disease other than heart failure that results in a life expectancy of <1 year (in the opinion of the investigator).
28. History or recurrent severe hypokalemia, potassium < 3.0 mg/dL.
29. Current enrollment or completion within 30 days of an investigational device or drug study.
30. Chronic alcohol or drug abuse or any condition that, in the investigator's opinion, will make the subject unlikely to fulfill the study requirements or complete the trial.
31. Any other clinical condition that might jeopardize subject safety during participation in this study or prevent the subject from adhering to the study protocol.
32. Unable or unwilling to follow guidelines of assigned diet group, including inability to purchase food.
33. Unable to participate in the comprehensive diet program, including biometric data acquisition and data entry.
34. The subject cannot currently be on a low-carb diet plan. 30-day washout would be required.
35. Patient has to have stable weight over the past 3 months (± 5% total body weight). If no weight was recorded in the past 3 months, will have 1 month lead in time for wash out.
36. Refusal to consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-05-19 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes in maximal exercise performance | baseline, 6 weeks, and end of the study (26 weeks)
  Participants will undergo VO2 max testing, conducted by trained professionals. VO2 max testing analyses will determine changes in maximal exercise performance

SECONDARY OUTCOMES:
Change in Cardiac Output (L/min) via cardiovascular magnetic resonance imaging (CMR) . | baseline, 6 weeks, and end of the study (26 weeks)
  Changes in cardiac output will be assessed via Cardiovascular magnetic resonance imagining conducted by trained professionals. MRI imaging analyses will determine cardiac function. The images will be analyzed by trained imaging professionals to determine overall change (L/min).
Change Stroke Volume(mL) via cardiovascular magnetic resonance imaging (CMR) | baseline, 6 weeks, and end of the study (26 weeks)
  Changes in stroke volume will be assessed via Cardiovascular magnetic resonance imagining conducted by trained professionals. MRI imaging analyses will determine cardiac function. The images will be analyzed by trained imaging professionals to determine change in stroke volume (mL).
Percent change in ejection fraction via cardiovascular magnetic resonance imaging (CMR) | baseline, 6 weeks, and end of the study (26 weeks)
  Percent changes in ejection fraction will be assessed via Cardiovascular magnetic resonance imagining conducted by trained professionals. MRI imaging analyses will determine cardiac function. The images will be analyzed by trained imaging professionals to determine change in Ejection Fraction(%).
Change in New York Heart Association (NYHA) class | baseline, 6 weeks, and end of the study (26 weeks)
  NYHA class will be determined by clinical examination by a qualified cardiovascular physician
Change in Quality of Life Questionnaire | baseline, 6 weeks, and end of the study (26 weeks)
  Participants will complete a quality of life questionnaire several times throughout the study. The questions are divided into three areas: Dyspnea, Fatigue and Emotional Function. The scores for each area are added up and divided by the number of questions. A 7-point scale is used for all areas where 1 is the best and 7 is the worst.
Metabolic Panel | baseline, 6 weeks, and end of the study (26 weeks)
  Changes in metabolic blood panel will be assessed at in lab visits (baseline, 6 weeks, and end of the study (26 weeks))
Lipid Panel | baseline, 6 weeks, and end of the study (26 weeks)
  Changes in lipid blood panel will be assessed at in lab visits (baseline, 6 weeks, and end of the study (26 weeks))
B-natriuretic peptide (BNP) | baseline, 6 weeks, and end of the study (26 weeks)
  Changes in BNP (pg/mL) will be assessed at in lab visits (baseline, 6 weeks, and end of the study (26 weeks)).
Continuous glucose/ketone monitor (CGM/CKM) | Up to ~ 26 weeks
  changes in daily glucose and ketone levels.

CONTACTS AND LOCATIONS:
Overall Officials: Yuchi Han, MD, MMSc, Principal Investigator — Ohio State University
Locations (1):
- The Ross Heart Hospital, Columbus, Ohio, United States